CLINICAL TRIAL: NCT02489643
Title: Role of an Individualized Medical Training in Improving Efficacy and Adherence to a 4-week Treatment With Calcipotriol and Betamethasone Dipropionate Gel for Mild-to-moderate Plaque Psoriasis
Brief Title: Individualized Medical Training and Calcipotriol and Betamethasone Dipropionate Gel in Plaque Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Giacomo Caldarola, MD, PhD, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11134/14
Record Dates: First submitted 2015-06-29; First posted 2015-07-03 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Receiving training (Experimental): Patients will be visited and receive information about the prescribed topical treatment according to the normal course and procedure of an outpatient visit at our institution. At the end of the visit, they will also receive practical instructions on dosages and application modalities of the topical therapy.
  Interventions: Procedure: Individualized practical training
- No-receiving training (No Intervention)

INTERVENTIONS:
Procedure: Individualized practical training
  Arms: Receiving training

SUMMARY:
The aim of the study will be to evaluate the impact of this individualized practical training on efficacy (evaluated by Psoriasis Area and Severity Index (PASI) and Body Surface Area (BSA) score performed by a physician blinded to the study groups) and adherence (calculated as days wherein gel was applied and as BSA/weight of gel applied rate) to a 4 week long treatment with dovobet gel. On the other hand, the investigators will evaluate in both groups as demographic (as sex, age, job,..) or disease (as severity, duration, impact of quality of life,..) characteristics influence the adherence to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of psoriasis will be maid mainly on clinical findings. If doubts, a skin sample will be obtained and evaluated by histopathological examination.

Exclusion Criteria:

* Patients with palmoplantar, scalp, inverse, erythrodermic, guttate, pustular psoriasis will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Efficacy as measured by PASI improvement | 1 month
Efficacy as measured by BSA improvement | 1 month

SECONDARY OUTCOMES:
Adherence as measured by days wherein gel was applied | 1 month
Adherence as measured by BSA/weight of gel applied rate | 1 month